CLINICAL TRIAL: NCT02234323
Title: An Open-Label, Multicenter Evaluation of the Safety and Efficacy of Recombinant Coagulation Factor VIII Fc Fusion Protein (rFVIIIFc; BIIB031) in the Prevention and Treatment of Bleeding in Previously Untreated Patients With Severe Hemophilia A
Brief Title: An Open Label Study to Determine the Safety and Efficacy of Replacement Factor VIII Protein (Known as rFVIIIFc) in Previously Untreated Males With Severe Hemophilia A
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bioverativ, a Sanofi company (Industry)
Collaborators: Swedish Orphan Biovitrum (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 997HA306; 2013-005512-10 (EudraCT Number)
Record Dates: First submitted 2014-08-29; First posted 2014-09-09 (Estimated); Results first posted 2020-08-13 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2022-03

CONDITIONS: Hemophilia A
Keywords: prophylaxis treatment; Hemophilia A; Hemophilia; episodic treatment
MeSH Terms: conditions — Hemophilia A | interventions — factor VIII-Fc fusion protein; Factor VIII

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- rFVIIIFc (Experimental): Participants were to receive rFVIIIFc as follows- Prophylaxis regimen (PR): rFVIIIFc 25-80 international units per kilogram (IU/kg), at 3- to 5-day intervals until participant reached greater than or equal to (>=) 50 exposure days (ED: 24-hour period in which >=1 injection/dose of rFVIIIFc was given), or study withdrawal/end of study. Adjustments to dose/dosing interval was done as needed by investigator; Treatment with an optional ER (Episodic regimen) can be initiated before PR at investigators discretion; ITI: rFVIIIFc 200 IU/kg, daily for participants who, after exposure to rFVIIIFc, had positive high titer inhibitor (>=5.00 Bethesda Units per milliliter [BU/mL]) or positive low titer inhibitor (>=0.60 and <5.00 BU/mL) and had poorly controlled bleeding despite increased rFVIIIFc doses, or required bypassing agent to treat bleeding.
  Interventions: Biological: rFVIIIFc

INTERVENTIONS:
Biological: rFVIIIFc — Administered as specified in arm description
  Other Names: Eloctate; BIIB031; efmoroctocog alfa; recombinant coagulation factor VIII Fc fusion protein; antihemophilic factor [recombinant]; Fc fusion protein

SUMMARY:
The primary objective of the study was to evaluate the safety of rFVIIIFc (BIIB031) in previously untreated participants (PUPs) with severe hemophilia A. The secondary objectives were to evaluate the efficacy of rFVIIIFc in the prevention and treatment of bleeding episodes in PUPs, to evaluate rFVIIIFc consumption for the prevention and treatment of bleeding episodes in PUPs, and to describe experience with the use of rFVIIIFc for immune tolerance induction (ITI) in participants with inhibitors.

ELIGIBILITY:
Key Inclusion Criteria:

* Ability of the participant's legally authorized representative (e.g. their parent or legal guardian) to understand the purpose and risks of the study and provide signed and dated informed consent and authorization to use confidential health information in accordance with national and local participant privacy regulations.
* Weight >=3.5 kg at the time of screening.
* Severe hemophilia A defined as less than (<) 1 IU/dL (<1%) endogenous FVIII documented in the medical record or as tested during the Screening Period.

Key Exclusion Criteria:

* Any exposure to blood components, factor VIII replacement products, including commercially available rFVIIIFc at any time prior to or during screening.
* History of positive inhibitor testing. A prior history of inhibitors was defined based on a patient's historical positive inhibitor test using the local laboratory Bethesda value for a positive inhibitor test (ie, equal to or above lower level of detection).
* History of hypersensitivity reactions associated with any rFVIIIFc administration.
* Other coagulation disorder(s) in addition to hemophilia A.
* Any concurrent clinically significant major disease that, in the opinion of the Investigator, would make the participant unsuitable for enrollment.
* Current systemic treatment with chemotherapy and/or other immunosuppressant drugs.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Max Age: 5 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 108 (Actual)
Dates: Start 2015-01-12 (Actual); Primary Completion 2019-09-23 (Actual); Study Completion 2019-09-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (69):
- United States (19):
  - Research Site, Little Rock, Arkansas
  - Research Site, Duarte, California
  - Research Site, Sacramento, California
  - Research Site, San Francisco, California
  - Research Site, Torrance, California
  - Research Site, Indianapolis, Indiana
  - Research Site, Louisville, Kentucky
  - Research Site, Brewer, Maine
  - Research Site, East Lansing, Michigan
  - Research Site, Minneapolis, Minnesota
  - Research Site, St Louis, Missouri
  - Research Site, Buffalo, New York
  - Research Site, New York, New York
  - Research Site, Rochester, New York
  - Research Site, Columbus, Ohio
  - Research Site, Portland, Oregon
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Dallas, Texas
  - Research Site, Milwaukee, Wisconsin
- Australia (4):
  - Research Site, Brisbane
  - Research Site, Parkville
  - Research Site, Perth
  - Research Site, Westmead
- Brazil (5):
  - Research Site, Campinas
  - Research Site, Canoas
  - Research Site, Ribeirão Preto
  - Research Site, Rio de Janeiro
  - Research Site, São Paulo
- Canada (3):
  - Research Site, Hamilton
  - Research Site, London
  - Research Site, Toronto
- France (7):
  - Research Site, Caen
  - Research Site, Le Kremlin-Bicêtre
  - Research Site, Lille
  - Research Site, Nantes
  - Research Site, Strasbourg
  - Research Site, Toulouse
  - Research Site, Tours
- Germany (5):
  - Research Site, Berlin
  - Research Site, Bonn
  - Research Site, Düsseldorf
  - Research Site, Frankfurt
  - Research Site, Hannover
- Research Site, Dublin, Ireland
- Italy (8):
  - Research Site, Vicenza, VI
  - Research Site, Bari
  - Research Site, Florence
  - Research Site, Genova
  - Research Site, Milan
  - Research Site, Napoli
  - Research Site, Padua
  - Research Site, Rome
- Netherlands (2):
  - Research Site, Leiden
  - Research Site, Utrecht
- New Zealand (2):
  - Research Site, Auckland
  - Research Site, Christchurch
- Poland (4):
  - Research Site, Gdansk
  - Research Site, Krakow
  - Research Site, Lublin
  - Research Site, Warsaw
- Spain (2):
  - Research Site, Barcelona
  - Research Site, Madrid
- Research Site, Stockholm, Sweden
- United Kingdom (6):
  - Research Site, Cambridge, Cambridgeshire
  - Research Site, Basingstoke, Hampshire
  - Research Site, Whitechapel, London
  - Research Site, Cardiff
  - Research Site, London
  - Research Site, Sheffield

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Carcao M, Schiavulli M, Kulkarni R, Rendo P, Foster M, Santagostino E, Casiano S, Konigs C. A post hoc analysis of previously untreated patients with severe hemophilia A who developed inhibitors in the PUPs A-LONG trial. Blood Adv. 2024 Mar 26;8(6):1494-1503. doi: 10.1182/bloodadvances.2023011475. PMID 38266154
- [Derived] Konigs C, Ozelo MC, Dunn A, Kulkarni R, Nolan B, Brown SA, Schiavulli M, Gunawardena S, Mukhopadhyay S, Jayawardene D, Winding B, Carcao M. First study of extended half-life rFVIIIFc in previously untreated patients with hemophilia A: PUPs A-LONG final results. Blood. 2022 Jun 30;139(26):3699-3707. doi: 10.1182/blood.2021013563. PMID 35421219

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 44 active centers in 13 countries between 12-Jan-2015 to 23-Sep-2019.
Pre-assignment Details: 110 participants screened, 108 enrolled, 103 received drug.
Groups:
- Recombinant Coagulation Factor VIII Fc Fusion Protein: Participants were to receive rFVIIIFc as follows -Prophylaxis regimen (PR): rFVIIIFc 25-80 international units per kilogram (IU/kg), at 3-5 day intervals until participant reached >= 50 exposure days (ED: 24-hour period in which >=1 injection/dose of rFVIIIFc was given), or study withdrawal/end of study. Adjustments to dose/dosing interval was done as needed by investigator; Treatment with an optional ER (Episodic regimen) can be initiated before PR at investigators discretion; ITI: rFVIIIFc 200 IU/kg, daily for participants who, after exposure to rFVIIIFc, had positive high titer inhibitor (>=5.00 Bethesda Units per milliliter [BU/mL]) or positive low titer inhibitor (>=0.60 and <5.00 BU/mL) and had poorly controlled bleeding despite increased rFVIIIFc doses, or required bypassing agent to treat bleeding.
Period: All Enrolled
Arm/Group | Recombinant Coagulation Factor VIII Fc Fusion Protein
Started | 108
Completed | 103 (These participants received at least one dose of study drug.)
Not Completed | 5
Not completed — Not Treated: Completed study in database | 2
Not completed — Not Treated:Consent withdrawn by subject | 2
Not completed — Not Treated: Exceeded lab value limit | 1
Period: All Treated
Arm/Group | Recombinant Coagulation Factor VIII Fc Fusion Protein
Started | 103
Episodic Treatment Regimen | 81 (Participants were treated in more than one regimen and counted in all categories wherever applicable)
Prophylactic Treatment Regimen | 89 (69 participants among the 81 who started in episodic regimen, switched to the prophylactic regimen.)
Immune Tolerance Induction (ITI) | 15 (1/81 on episodic and 14/89 on prophylactic regimen had inhibitors and were switched directly to ITI.)
Completed | 85
Not Completed | 18
Not completed — Death | 1
Not completed — Physician Decision | 5
Not completed — Lack of Efficacy | 3
Not completed — Exceeded lab value limit | 2
Not completed — Other | 7

BASELINE CHARACTERISTICS:
Population: The safety analysis set was defined as all participants who received at least 1 dose of rFVIIIFc.
Groups:
- Recombinant Coagulation Factor VIII Fc Fusion Protein: Participants were to receive rFVIIIFc as follows -PR: rFVIIIFc 25-80 IU/kg, at 3- to 5-day intervals until participant reached >= 50 exposure days (ED: 24-hour period in which >=1 injection/dose of rFVIIIFc was given), or study withdrawal/end of study. Adjustments to dose/dosing interval was done as needed by investigator; Treatment with an optional ER can be initiated before PR at investigators discretion; ITI: rFVIIIFc 200 IU/kg, daily for participants who, after exposure to rFVIIIFc, had positive high titer inhibitor (>=5.00 BU/mL) or positive low titer inhibitor (>=0.60 and <5.00 BU/mL) and had poorly controlled bleeding despite increased rFVIIIFc doses, or required bypassing agent to treat bleeding.
Arm/Group | Recombinant Coagulation Factor VIII Fc Fusion Protein
Number analyzed (Participants) | 103
Age, Continuous [Median (Full Range); unit: years] | 0.58 [0.02 to 4.00]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 103
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 79
  Black or African-American | 2
  Asian | 5
  Native Hawaiian or other Pacific Islander | 2
  Not reported due to confidentiality regulations | 4
  Other | 11

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Confirmed Inhibitor Development as Measured by the Nijmegen-Modified Bethesda Assay
Description: A positive/confirmed inhibitor result occurs when a participant has a value >=0.6 BU/mL by central laboratory testing using Nijmegen-modified Bethesda assay, that is confirmed on re-testing of a separate sample collected >=2 weeks after the initial sample. Confirmed inhibitor development was based on all participants who had reached >=10 EDs and had >=1 inhibitor test performed at or beyond this milestone or who had an inhibitor. Exposure day (ED) is a 24-hour period in which participant received >=1 dose of rFVIIIFc injections. Participants who did not develop an inhibitor but reached the milestone number of EDs were included in the denominator during calculation of percentage. Additionally, any participant who developed an inhibitor following the initial rFVIIIFc administration was included in the numerator and denominator during calculation of percentage.
Time Frame: Up to 3 years
Population: Safety analysis set participants who 1) reached >=10 EDs and had >=1 inhibitor test performed at >=10 EDs or who had inhibitor or 2) did not develop inhibitor but reached >=10 EDs or 3) developed an inhibitor following the initial rFVIIIFc administration.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Recombinant Coagulation Factor VIII Fc Fusion Protein: Participants were to receive rFVIIIFc as follows -PR (Prophylaxis regimen): rFVIIIFc 25-80 IU/kg, at 3- to 5-day intervals until participant reached >= 50 exposure days (ED: 24-hour period in which >=1 injection/dose of rFVIIIFc was given), or study withdrawal/end of study. Adjustments to dose/dosing interval was done as needed by investigator; Treatment with an optional ER can be initiated before PR at investigators discretion; ITI: rFVIIIFc 200 IU/kg, daily for participants who, after exposure to rFVIIIFc, had positive high titer inhibitor (>=5.00 BU/mL) or positive low titer inhibitor (>=0.60 and <5.00 BU/mL) and had poorly controlled bleeding despite increased rFVIIIFc doses, or required bypassing agent to treat bleeding.
Arm/Group | Recombinant Coagulation Factor VIII Fc Fusion Protein
Number analyzed (Participants) | 90
percentage of participants | 31.11 [21.77 to 41.74]

2. Secondary Outcome: Annualized Number of Bleeding Episodes (Spontaneous and Traumatic) Per Participant (Annualized Bleeding Rate [ABR])
Description: ABR was annualized number of bleeding episodes during efficacy period (EP) per participant annualized to a 1-year interval of time. Bleeding episodes were classified as spontaneous if parent/caregiver/participant records bleeding event when there is no known contributing factor such as definite trauma or antecedent "strenuous" activity and as traumatic when there is known reason for bleed. ABR=(Number of bleeding episodes during EP divided by total number of days during EP)*365.25. EP was sum of all intervals of time during which participants were treated with rFVIIIFc per treatment regimens of study excluding surgical/rehabilitation periods and large injection intervals (greater than [>]28 days). Participants were included in summary of more than 1 treatment regimen if their regimen changed during study.
Time Frame: Up to 3 years
Population: Analysis performed on Full Analysis Set (FAS) participants within the EP. FAS included all enrolled participants with >=1 dose of study treatment. Here, number analyzed signifies number of FAS participants analyzed in each treatment regimen.
Measure: Median (Full Range); unit: episodes per participant per year
Arm/Group | Recombinant Coagulation Factor VIII Fc Fusion Protein
Number analyzed (Participants) | 101
episodes per participant per year
  Episodic Treatment: number analyzed (Participants) | 81
  Episodic Treatment | 2.24 [0.0 to 39.8]
  Prophylaxis Treatment: number analyzed (Participants) | 89
  Prophylaxis Treatment | 1.49 [0.0 to 18.7]
  ITI Treatment: number analyzed (Participants) | 15
  ITI Treatment | 0.00 [0.0 to 6.6]

3. Secondary Outcome: Annualized Number of Spontaneous Joint Bleeding Episodes
Description: Bleeding episodes were classified as spontaneous if parent/caregiver/participant records a bleeding event when there was no known contributing factor such as a definite trauma or antecedent "strenuous" activity. Annualized spontaneous joint bleeding episodes = (Total number of spontaneous joint bleeding episodes during EP divided by total number of days during EP)*365.25. EP reflects sum of all intervals of time during which participants were treated with rFVIIIFc per treatment regimen excluding major and minor surgical/rehabilitation periods and large injection intervals (> 28 days). Bleeding episodes were summarized by treatment regimen. Participants were included in summary of more than 1 treatment regimen if their regimen changed during study.
Time Frame: Up to 3 years
Population: Analysis was performed on FAS which included participants within EP. Here, number analyzed signifies number of FAS participants who were analyzed in each treatment regimen.
Measure: Median (Inter-Quartile Range); unit: episodes per participant per year
Arm/Group | Recombinant Coagulation Factor VIII Fc Fusion Protein
Number analyzed (Participants) | 101
episodes per participant per year
  Episodic Treatment: number analyzed (Participants) | 81
  Episodic Treatment | 0.00 [0.0 to 0.0]
  Prophylaxis Treatment: number analyzed (Participants) | 89
  Prophylaxis Treatment | 0.00 [0.0 to 0.0]
  ITI Treatment: number analyzed (Participants) | 15
  ITI Treatment | 0.00 [0.0 to 0.0]

4. Secondary Outcome: Number of rFVIIIFc Injections With Excellent or Good, Moderate or None Treatment Response Assessed Using a 4-Point Scale
Description: Using e-diary, each participant's parent/caregiver rated treatment response to any bleeding episode at approximately 8-12 hours from time of injection and prior to additional doses of rFVIIIFc given for same bleeding episodes, using 4-point scale: 1=Excellent: abrupt pain relief and/or improvement in signs of bleeding within approximately 8 hour after initial injection; 2=Good: definite pain relief and/or improvement in signs of bleeding within approximately 8 hour after injection, but possibly requiring more than 1 injection after 24-48 hour for complete resolution; 3=Moderate: Probable/slight beneficial effect within 8 hour after initial injection and requires more than 1 injection and 4=None: No improvement or condition worsens within approximately 8 hour after initial injection. Participants included in more than 1 treatment regimen if their regimen changed during study.
Time Frame: Up to 3 years
Population: Analysis performed on FAS participants within the EP and based on all injections. Here, number analyzed signifies number of responses to injections reported for each treatment regimen.
Measure: Count of Units; unit: responses to injections
Units Other Than Participants: responses to injections
Arm/Group | Recombinant Coagulation Factor VIII Fc Fusion Protein
Number analyzed (Participants) | 101
Number analyzed (responses to injections) | 579
responses to injections
  Episodic Regimen: number analyzed (Participants) | 81
  Episodic Regimen: number analyzed (responses to injections) | 238
  Episodic Regimen: Excellent or Good | 102
  Episodic Regimen: Moderate | 16
  Episodic Regimen: None | 2
  Episodic Regimen: Response not provided | 118
  Prophylaxis Regimen: number analyzed (Participants) | 89
  Prophylaxis Regimen: number analyzed (responses to injections) | 293
  Prophylaxis Regimen: Excellent or Good | 163
  Prophylaxis Regimen: Moderate | 27
  Prophylaxis Regimen: None | 14
  Prophylaxis Regimen: Response not provided | 89
  ITI Regimen: number analyzed (Participants) | 15
  ITI Regimen: number analyzed (responses to injections) | 48
  ITI Regimen: Excellent or Good | 20
  ITI Regimen: Moderate | 14
  ITI Regimen: None | 3
  ITI Regimen: Response not provided | 11

5. Secondary Outcome: Total Number of Exposure Days (EDs)
Description: An ED was defined as a 24-hour period in which a participant received one or more doses of rFVIIIFc injections, with the time of the first injection of rFVIIIFc defined as the start of the ED. Participants who did not have a particular injection type were counted as having zero injections for that type.
Time Frame: Up to 3 years
Population: Analysis performed on safety analysis set.
Measure: Median (Full Range); unit: days
Arm/Group | Recombinant Coagulation Factor VIII Fc Fusion Protein
Number analyzed (Participants) | 103
days | 100.0 [0 to 649]

6. Secondary Outcome: Total Annualized rFVIIIFc Consumption Per Participant for the Prevention and Treatment of Bleeding Episodes
Description: Total annualized rFVIIIFc consumption (in IU/kg) was calculated for each participant as: Annualized consumption = (Total IU/kg of rFVIIIFc during EP divided by total number of days during EP)*365.25. EP reflects the sum of all intervals of time during which participants are treated with rFVIIIFc according to the treatment regimens of the study excluding surgical/rehabilitation periods and large injection intervals (>28 days). Participants were included in summary of more than 1 treatment regimen if their regimen changed during study.
Time Frame: Up to 3 years
Population: Analysis performed on FAS participants within the EP. Here, number analyzed signifies number of FAS participants who were analyzed in each treatment regimen.
Measure: Median (Full Range); unit: IU per kilogram per participant per year
Arm/Group | Recombinant Coagulation Factor VIII Fc Fusion Protein
Number analyzed (Participants) | 101
IU per kilogram per participant per year
  Episodic Treatment: number analyzed (Participants) | 81
  Episodic Treatment | 197.6 [0 to 3177]
  Prophylaxis Treatment: number analyzed (Participants) | 89
  Prophylaxis Treatment | 5384.4 [0 to 40126]
  ITI Treatment: number analyzed (Participants) | 15
  ITI Treatment | 67310.0 [33323 to 78871]

7. Secondary Outcome: Number of Injections of rFVIIIFc Required to Resolve a Bleeding Episode
Description: Number of Injections of rFVIIIFc required to resolve a bleeding episode during EP were reported. EP reflects the sum of all intervals of time during which participants were treated with rFVIIIFc according to the treatment regimens of the study excluding surgical/rehabilitation periods and large injection intervals (>28 days). All injections given from the initial sign of a bleed, until the last date/time within the bleed window were counted. Participants were included in summary of more than 1 treatment regimen if their regimen changed during study.
Time Frame: Up to 3 years
Population: as for outcome 6
Measure: Median (Full Range); unit: injections
Arm/Group | Recombinant Coagulation Factor VIII Fc Fusion Protein
Number analyzed (Participants) | 101
injections
  Episodic Treatment: number analyzed (Participants) | 81
  Episodic Treatment | 1.0 [1 to 13]
  Prophylaxis Treatment: number analyzed (Participants) | 89
  Prophylaxis Treatment | 1.0 [1 to 7]
  ITI Treatment: number analyzed (Participants) | 15
  ITI Treatment | 1.0 [1 to 22]

8. Secondary Outcome: Average Dose Per Injection of rFVIIIFc Required to Resolve a Bleeding Episode
Description: The average dose of rFVIIIFc per injection per bleeding episode was calculated as the average of all doses (IU/kg) administered to treat the bleeding episode during EP. EP begins with the first treatment regimen dose of rFVIIIFc and ends with the last dose (regardless of the reason for dosing). Surgery/rehabilitation periods were not included in the EP. Participants were included in summary of more than 1 treatment regimen if their regimen changed during study.
Time Frame: Up to 3 years
Population: as for outcome 6
Measure: Median (Full Range); unit: IU/kg
Arm/Group | Recombinant Coagulation Factor VIII Fc Fusion Protein
Number analyzed (Participants) | 101
IU/kg
  Episodic Treatment: number analyzed (Participants) | 81
  Episodic Treatment | 45.45 [19.2 to 106.0]
  Prophylaxis Treatment: number analyzed (Participants) | 89
  Prophylaxis Treatment | 48.08 [17.9 to 144.0]
  ITI Treatment: number analyzed (Participants) | 15
  ITI Treatment | 189.44 [76.9 to 250.0]

9. Secondary Outcome: Change From Baseline in rFVIIIFc Incremental Recovery (IR)
Description: Blood samples were taken at trough (predose) and Cmax (maximum concentration) for assessment of incremental recovery, measured by the one-stage clotting assay. IR (International Units per deciliter [IU/dL] per IU/kg) = (Cmax for FVIII activity - Pre-dose FVIII activity) (IU/dL) divided by actual dose (IU/kg), where Cmax (maximum concentration) is 30-minute FVIII activity post-dose and FVIII activity less than (<)0.5 IU/dL was set to 0 IU/dL for calculation of IR.
Time Frame: Baseline, Weeks 12, 24, 36, 48, 60, 72, 84, 96, 108 and 120
Population: Analysis performed on FAS participants within the EP. Here number analyzed signifies number of FAS participants with available data for each visit.
Measure: Median (Inter-Quartile Range); unit: IU/dL per IU/kg
Groups:
- Recombinant Coagulation Factor VIII Fc Fusion Protein: Participants were to receive rFVIIIFc as follows -PR: rFVIIIFc 25-80 IU/kg, at 3- to 5-day intervals until participant reached >= 50 exposure days (ED: 24-hour period in which >=1 injection/dose of rFVIIIFc was given), or study withdrawal/end of study. Adjustments to dose/dosing interval was done as needed by investigator; Treatment with an optional ER (Episodic regimen) can be initiated before PR at investigators discretion; ITI: rFVIIIFc 200 IU/kg, daily for participants who, after exposure to rFVIIIFc, had positive high titer inhibitor (>=5.00 BU/mL) or positive low titer inhibitor (>=0.60 and <5.00 BU/mL) and had poorly controlled bleeding despite increased rFVIIIFc doses, or required bypassing agent to treat bleeding.
Arm/Group | Recombinant Coagulation Factor VIII Fc Fusion Protein
Number analyzed (Participants) | 101
IU/dL per IU/kg
  Change at Week 12: number analyzed (Participants) | 35
  Change at Week 12 | -0.5 [-1.26 to -0.26]
  Change at Week 24: number analyzed (Participants) | 34
  Change at Week 24 | -0.7 [-1.50 to 0.05]
  Change at Week 36: number analyzed (Participants) | 39
  Change at Week 36 | -0.4 [-1.06 to 0.27]
  Change at Week 48: number analyzed (Participants) | 37
  Change at Week 48 | -0.5 [-1.09 to -0.05]
  Change at Week 60: number analyzed (Participants) | 25
  Change at Week 60 | -0.4 [-1.06 to 0.04]
  Change at Week 72: number analyzed (Participants) | 21
  Change at Week 72 | -0.8 [-1.10 to -0.24]
  Change at Week 84: number analyzed (Participants) | 15
  Change at Week 84 | -0.6 [-1.55 to 0.01]
  Change at Week 96: number analyzed (Participants) | 7
  Change at Week 96 | -0.6 [-1.21 to -0.34]
  Change at Week 108: number analyzed (Participants) | 2
  Change at Week 108 | -1.5 [-2.68 to -0.31]
  Change at Week 120: number analyzed (Participants) | 1
  Change at Week 120 | -0.6 [-0.6 to -0.6]

10. Secondary Outcome: Number of Participants With Response to Immune Tolerance Induction (ITI)
Description: Complete Success was defined as meeting all of the following criteria: Negative inhibitor titers in 2 consecutive determinations at least 4 weeks apart; IR >=66% of baseline in 2 consecutive determinations at least 4 weeks apart; Half life >=6 hours. Partial Success was defined as meeting the first criteria for complete success and one of the other 2 after 33 months of ITI.
Time Frame: Up to 3 years
Population: Analysis performed on ITI analysis set which was defined as all participants who consented to and initiated the ITI sub-study.
Measure: Count of Participants; unit: Participants
Arm/Group | Recombinant Coagulation Factor VIII Fc Fusion Protein
Number analyzed (Participants) | 15
Participants
  Complete Success | 5
  Partial Success | 2
  Early Withdrawal | 3
  ITI Ongoing at end of Study | 5

ADVERSE EVENTS:
Time Frame: All Adverse Events (AEs) were collected from signature of the informed consent form up to end of the study (up to 3 years) regardless of seriousness or relationship to investigational product.
Description: Reported AEs are treatment-emergent AEs i.e. AE that was present prior to receiving first injection of rFVIIIFc and subsequently worsened in severity, or was not present prior to receiving first injection but subsequently appeared before last visit/follow-up call, whichever came later. Analysis performed on safety analysis set.
Arm/Group | Recombinant Coagulation Factor VIII Fc Fusion Protein
All-Cause Mortality (participants affected / at risk) | 1/103
Serious Adverse Events (participants affected / at risk) | 60/103
Other Adverse Events (participants affected / at risk) | 85/103
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Recombinant Coagulation Factor VIII Fc Fusion Protein (N=103)
Factor viii inhibition (Blood and lymphatic system disorders) | 28 (29)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Spontaneous haematoma (Blood and lymphatic system disorders) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1)
Tongue haemorrhage (Gastrointestinal disorders) | 1 (1)
Device related thrombosis (General disorders) | 1 (1)
Pyrexia (General disorders) | 4 (4)
Bacterial sepsis (Infections and infestations) | 1 (1)
Gastroenteritis norovirus (Infections and infestations) | 1 (1)
Haematoma infection (Infections and infestations) | 1 (1)
Meningitis aseptic (Infections and infestations) | 1 (1)
Parainfluenzae virus infection (Infections and infestations) | 2 (2)
Pneumonia (Infections and infestations) | 2 (2)
Rotavirus infection (Infections and infestations) | 1 (1)
Staphylococcal bacteraemia (Infections and infestations) | 1 (2)
Staphylococcal infection (Infections and infestations) | 2 (2)
Staphylococcal skin infection (Infections and infestations) | 1 (1)
Vascular device infection (Infections and infestations) | 2 (3)
Viral infection (Infections and infestations) | 2 (2)
Viral upper respiratory tract infection (Infections and infestations) | 2 (2)
Concussion (Injury, poisoning and procedural complications) | 1 (4)
Contusion (Injury, poisoning and procedural complications) | 1 (1)
Craniocerebral injury (Injury, poisoning and procedural complications) | 2 (2)
Facial bones fracture (Injury, poisoning and procedural complications) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 11 (19)
Head injury (Injury, poisoning and procedural complications) | 8 (13)
Palate injury (Injury, poisoning and procedural complications) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1)
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 (1)
Vascular access site haematoma (Injury, poisoning and procedural complications) | 1 (1)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 2 (2)
Haematoma muscle (Musculoskeletal and connective tissue disorders) | 1 (1)
Soft tissue haemorrhage (Musculoskeletal and connective tissue disorders) | 1 (1)
Febrile convulsion (Nervous system disorders) | 2 (2)
Haemorrhage intracranial (Nervous system disorders) | 2 (2)
Intraventricular haemorrhage (Nervous system disorders) | 1 (1)
Device issue (Product Issues) | 1 (1)
Mental status changes (Psychiatric disorders) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Arteriovenous fistula operation (Surgical and medical procedures) | 1 (1)
Central venous catheter removal (Surgical and medical procedures) | 1 (1)
Central venous catheterisation (Surgical and medical procedures) | 26 (30)
Ventriculo-peritoneal shunt (Surgical and medical procedures) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1)
Haematoma (Vascular disorders) | 3 (3)
Poor venous access (Vascular disorders) | 3 (3)
Subgaleal haematoma (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Recombinant Coagulation Factor VIII Fc Fusion Protein (N=103)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 10 (10)
Constipation (Gastrointestinal disorders) | 9 (9)
Diarrhoea (Gastrointestinal disorders) | 18 (23)
Teething (Gastrointestinal disorders) | 12 (23)
Vomiting (Gastrointestinal disorders) | 19 (20)
Pyrexia (General disorders) | 31 (47)
Conjunctivitis (Infections and infestations) | 8 (8)
Ear infection (Infections and infestations) | 19 (28)
Gastroenteritis (Infections and infestations) | 7 (7)
Hand-foot-and-mouth disease (Infections and infestations) | 6 (6)
Influenza (Infections and infestations) | 10 (14)
Nasopharyngitis (Infections and infestations) | 31 (54)
Otitis media (Infections and infestations) | 10 (11)
Rhinitis (Infections and infestations) | 7 (11)
Upper respiratory tract infection (Infections and infestations) | 28 (41)
Varicella (Infections and infestations) | 6 (6)
Viral infection (Infections and infestations) | 17 (32)
Viral upper respiratory tract infection (Infections and infestations) | 11 (27)
Contusion (Injury, poisoning and procedural complications) | 9 (16)
Fall (Injury, poisoning and procedural complications) | 52 (146)
Head injury (Injury, poisoning and procedural complications) | 28 (63)
Limb injury (Injury, poisoning and procedural complications) | 8 (9)
Lip injury (Injury, poisoning and procedural complications) | 6 (6)
Mouth injury (Injury, poisoning and procedural complications) | 9 (10)
Skin abrasion (Injury, poisoning and procedural complications) | 7 (19)
Skin laceration (Injury, poisoning and procedural complications) | 9 (13)
Vaccination complication (Injury, poisoning and procedural complications) | 6 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 13 (20)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 9 (9)
Eczema (Skin and subcutaneous tissue disorders) | 6 (9)
Rash (Skin and subcutaneous tissue disorders) | 10 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2018-02-12): https://cdn.clinicaltrials.gov/large-docs/23/NCT02234323/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-30): https://cdn.clinicaltrials.gov/large-docs/23/NCT02234323/SAP_001.pdf